CLINICAL TRIAL: NCT02373696
Title: Prediction of Chronic Pain in the Asian Population- Comprehensive Programme Encompassing Dynamic Psychophysical Tests and Genetic Screening to Determine and Prevent Persistent Post-caesarean Pain
Brief Title: Chronic Pain Dynamic Psychophysical Tests and Genetic Screening
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2010/160/D
Record Dates: First submitted 2015-02-22; First posted 2015-02-27 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: Pain; Caesarean section
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sampling
Oversight: Data Monitoring Committee: No

SUMMARY:
Incidence and risk factors for persistent post surgical pain after Caesarean section are investigated. Demographic, psychophysical testing and genetic screening factors are performed in the perioperative period. Phone survey is performed to investigate the incidence of persistent post surgical pain after Caesarean section.

DETAILED DESCRIPTION:
Persistent post surgical pain after Caesarean section may lead to functional limitation and pain during activities of daily living. Demographic factors, psychophysical factors (mechanical temporal summation, diffuse noxious inhibitory control, state trait anxiety inventory) and genetic screening are used to predict the association with persistent post surgical pain. Phone survey follow up is performed to investigate the incidence of persistent post surgical pain and functional limitations due to pain experienced.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing spinal anaesthesia for Caesarean section

Exclusion Criteria:

* Failed spinal anaesthesia, Unable to perform psychophysical testing.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing spinal anaesthesia for Caesarean section
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2010-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Persistent Postsurgical Pain | 12 weeks
  Pain experienced in the lower abdominal region and surgical area after Caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore, Singapore